CLINICAL TRIAL: NCT04368377
Title: Platelet Inhibition With GP IIb/IIIa Inhibitor in Critically Ill Patients With Coronavirus Disease 2019 (COVID-19). A Compassionate Use Protocol
Brief Title: Enhanced Platelet Inhibition in Critically Ill Patients With COVID-19
Acronym: PIC-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Fondazione "Un Cuore per Milano" - a no profit foundation (Unknown)
Responsible Party: Principal Investigator, Pierachille Santus, MD, PhD, Professor of Respiratory Medicine, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18275/2020
Record Dates: First submitted 2020-04-23; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Pneumonia, Viral; Corona Virus Infection; Respiratory Failure; Embolism and Thrombosis
Keywords: Covid-19; Pneumonia; Respiratory failure; Platelet inhibition; GP IIb/IIIa inhibitor; Thrombosis; Platelet disfunction
MeSH Terms: conditions — Pneumonia, Viral; Coronavirus Infections; Respiratory Insufficiency; Embolism and Thrombosis; COVID-19; Pneumonia; Thrombosis | interventions — Tirofiban; Clopidogrel; Aspirin; Fondaparinux

STUDY DESIGN:
Intervention Model Description: Compassionate-use, proof of concept, interventional, prospective,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tirofiban (Experimental): 1. Patients will receive 25 microgram per kilogram of body weight tirofiban as bolus IV injection (3 minutes) followed by continuous infusion at a rate of 0.15 microgram/kg/minute for 48 hours.
  2. Patients will receive acetylsalicylic acid 250 mg IV before starting tirofiban, and this will be continued at a dose of 75 mg daily for 30 days.
  3. Patients will receive a loading dose of clopidogrel 300 mg PO, followed by 75 mg daily for 30 days
  4. Patents will receive concurrent fondaparinux 2.5 mg s/c per day for the duration of the hospital stay
  Interventions: Drug: Tirofiban Injection; Drug: Clopidogrel; Drug: Acetylsalicylic acid; Drug: Fondaparinux

INTERVENTIONS:
Drug: Tirofiban Injection — Patients will receive 25 microgram per kilogram of body weight tirofiban as bolus IV injection (3 minutes) followed by continuous infusion at a rate of 0,15 microgram/kg//minute for 48 hours.
  Other Names: Ibisqus; Agrastat
Drug: Clopidogrel — Patients will receive a loading dose of clopidogrel 300 mg PO, followed by 75mg daily for 30 days
  Other Names: Plavix
Drug: Acetylsalicylic acid — Patients will receive acetylsalicylic acid 250 mg IV before starting tirofiban, and this will be continued at a dose of 75mg daily for 30 days.
  Other Names: Cardirene
Drug: Fondaparinux — Patients will receive concurrent fondaparinux 2.5mg s/c per day for the duration of the in hospital stay
  Other Names: Arixtra

SUMMARY:
This is a compassionate use, proof of concept, phase IIb, prospective, interventional, pilot study in which the investigators will evaluate the effects of compassionate-use treatment with IV tirofiban 25 mcg/kg, associated with acetylsalicylic acid IV, clopidogrel PO and fondaparinux 2.5 mg s/c, in patients affected by severe respiratory failure in Covid-19 associated pneumonia who underwent treatment with continuous positive airway pressure (CPAP).

DETAILED DESCRIPTION:
It is a investigator-initiated, compassionate use, prospective, phase 2b, non randomized, open-label, proof of concept study in which the investigators will evaluate the effects of compassionate-use treatment with IV tirofiban, associated with acetylsalicylic acid PO, clopidogrel PO and fondaparinux 2.5 mg s/c, in patients affected by severe respiratory failure in Covid-19 associated pneumonia who underwent treatment with continuous positive airway pressure (CPAP).

Patients will be treated with:

1. 25 microgram per kilogram of body weight tirofiban as bolus IV injection (3 minutes) followed by continuous infusion at a rate of 0,15 microgram/kg/minute for 48 hours.
2. acetylsalicylic acid 250 mg IV before starting tirofiban, and this will be continued at a dose of 75mg daily for 30 days.
3. a loading dose of clopidogrel 300 mg PO, followed by 75mg daily for 30 days
4. concurrent fondaparinux 2.5 mg s/c per day for the duration of the in hospital stay.

1) Demographics, body mass index, comorbidities, SOFA score, APACHE II score, Glasgow Coma Scale will be assessed the day the patient is admitted to the IRCU.

2) Blood gas analysis parameters (PaO2, PaCO2, HCO3-, lactates, SaO2, pH), Alveolar-arterial gradient, P/F ratio, respiratory rate, arterial blood pressure, heart rate and Chest X ray or Chest CT scan will be collected at admittance following the standard operating procedures of the IRCU for COVID-19 patients. The same measurement as detailed in 2) will be repeated 1 hour before and 1, 24, 48 and 168 hours after the loading bolus of tirofiban.

Moreover, at admittance, participating patients will undergo a complete blood count, serum dosage of: creatinine, blood urea nitrogen (BUN), procalcitonin, c-reactive protein, Prothrombin Time (PT), Partial Thromboplastin Time (PTT), D-Dimer, fibrinogen, bilirubin, lactate dehydrogenase (LDH), aspartate transaminase (AST). The same assessment will be repeated the same morning and 24, 48 and 168 hours after the loading dose of tirofiban.

During hospital stay patients will receive continuous vital sign monitoring including: electrocardiogram tracing, blood arterial pressure, peripheral oxygen saturation and heart rate. Neurological status, signs of active bleeding or the occurrence of adverse effects will be monitored during the whole hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed SARS-CoV-2-related pneumonia, defined as positive nasal swab for SARS-CoV-2 infection or positive IgM serum title. A laboratory confirmed diagnosis must be associated with a clinically confirmed COVID-19 pneumonia, with a history of fever ≥ 3 days and multiple pulmonary infiltrates at the chest X-Ray
* Acute de novo severe hypoxic respiratory failure, defined by means of arterial blood gas analysis performed in room air showing severe hypoxemia with an arterial partial pressure of oxygen (PaO2) to fraction of inspired oxygen (FiO2) ratio < 250 (according to the Berlin 2012 acute respiratory distress syndrome - ARDS - definition), requiring CPAP respiratory support
* D-Dimer value ≥ 3 times the upper level of normal of the laboratory

Exclusion Criteria:

* Ongoing bleeding or bleeding diathesis, contraindications for anticoagulation or increased bleeding risk or history of bleeding in the last eight weeks
* Previous stroke or transient ischemic attack or any intracranial pathology in the last six months, major surgery or trauma within the previous six weeks
* Laboratory confirmed Laboratory confirmed Glucose 6-Phosphate Dehydrogenase (G6PDH) deficiency.
* Confirmed or suspected pregnancy or patients in childbearing age.
* Previous known adverse effects or intolerance to the study drugs
* Ongoing septic shock. Septic shock will be defined as the concomitant presence of sepsis (life-threatening organ dysfunction caused by a dysregulated host response to infection with a Sequential [Sepsis-related] Organ Failure Assessment (SOFA) score of 2 points or more) and need for vasopressors to maintain a mean arterial pressure of 65 mm Hg or greater and a serum lactate level greater than 2 mmol/L (>18 mg/dL) in the absence of hypovolemia.
* Need for surgery during hospitalization
* Elevated risk of in hospital fall
* Glasgow Coma Scale <15
* Confirmed diagnosis of dementia or mental disability that jeopardizes the comprehension of the study protocol
* Inability to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
P/F ratio | At baseline and 24, 48 and 168 hours after treatment initiation
  Change in ratio between partial pressure of oxygen in arterial blood, measured by means of arterial blood gas analysis, and inspired oxygen fraction at baseline and after study treatment
PaO2 difference | At baseline and 24, 48 and 168 hours after treatment initiation
  Change in partial pressure of oxygen in arterial blood, measured by means of arterial blood gas analysis, at baseline and after study treatment
A-a O2 difference | At baseline and 24, 48 and 168 hours after treatment initiation
  Change in alveolar-arterial gradient of oxygen at baseline and after study treatment. Arterial alveolar gradient will be calculated using the following parameters derived from arterial blood gas analysis: partial pressure of oxygen in arterial blood and partial pressure of carbon dioxide in arterial blood.

SECONDARY OUTCOMES:
CPAP duration | From the first day of study drugs administration (T0) until day 7 post study drugs administration
  Number of days on continuous positive end expiratory pressure (CPAP)
In-hospital change in intensity of the respiratory support | At baseline and 72 and 168 hours after treatment initiation
  Difference in intensity of the respiratory support (non invasive mechanical ventilation, CPAP, high flow nasal cannula (HFNC), Venturi Mask, nasal cannula, from higher to lower intensity, respectively) employed at baseline and at 72 and 168 hours after study treatment initiation
PaCO2 difference | At baseline and 24, 48 and 168 hours after treatment initiation
  Difference in partial pressure of carbon dioxide in arterial blood, measured by means of arterial blood gas analysis, at baseline and after study treatment
HCO3- difference | At baseline and 24, 48 and 168 hours after treatment initiation
  Difference in concentration of bicarbonate in arterial blood, measured by means of arterial blood gas analysis, at baseline and after study treatment
Lactate difference | At baseline and 24, 48 and 168 hours after treatment initiation
  Difference in concentration of lactate in arterial blood, measured by means of arterial blood gas analysis, at baseline and after study treatment
Hb difference | At baseline and 24, 48 and 168 hours after treatment initiation
  Difference in hemoglobin concentration in blood samples, measured by means of blood chemistry test, at baseline and after study treatment.
Plt difference | At baseline and 24, 48 and 168 hours after treatment initiation
  Difference in platelet concentration in blood samples, measured by means of blood chemistry test, at baseline and after study treatment.
Adverse effects | From the first day of study drugs administration until day 30 post study drugs administration
  Any major or minor adverse effect occuring during and after the administration of the study drug (e.g. bleeding)

CONTACTS AND LOCATIONS:
Locations (1):
- L. Sacco Hospital, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773